CLINICAL TRIAL: NCT05914415
Title: The Effect of Preoperative Structured Education Given to Patients Undergoing Mastectomy Surgery on the Quality of Post-operative Recovery
Brief Title: The Effect of Preoperative Education on Postoperative Healing Quality in Patients With Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EH2023SBU
Record Dates: First submitted 2022-08-26; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2022-08

CONDITIONS: Mastectomy; Lymphedema; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): standard preoperative training
  Interventions: Other: Supportive care and education before surgery
- Experimental (Experimental): structured training app
  Interventions: Other: Supportive care and education before surgery

INTERVENTIONS:
Other: Supportive care and education before surgery — we will give supportive and informative education before surgery in order to increase patient' recovery rates

SUMMARY:
Breast cancer is one of the most common types of cancer today. Treatment is planned depending on various factors. The most common treatment option is surgery. Mastectomy is a type of surgery in which the entire breast is removed. Tumorous tissue is removed with mastectomy, and cancer is treated, but after the intervention, physiological, psychological and social problems may occur in individuals in the acute and chronic periods. By providing pre-operative education, complications in the postoperative period can be reduced and the patient's compliance with the treatment can be ensured. It is stated in the studies that the training given by the nurses with different methods before the surgery reduces the anxiety, pain level and increases the comfort of the patients. No study was found in which the preoperative structured education given to patients scheduled for mastectomy was evaluated with the Postoperative Healing Quality Scale. The study is planned to be conducted as a randomized controlled experimental study and the patients who applied to Bakırköy Dr.Sadi Konuk Training and Research Hospital General Surgery Clinic for mastectomy constitute the research population. The sample is planned to consist of 70 patients, including 35 control and 35 experimental groups. In the structured training program in the research, both face-to-face information will be given to the patients and a written training booklet will be used. Patient Diagnosis Form, Recovery Quality Scale will be used to collect data. Through the data obtained, it will be evaluated whether the education given to the patients who are planned for mastectomy has an effect on the quality of recovery in the early postoperative period. It is thought that this study will reveal the benefits of preoperative education, increase the health care satisfaction of the patients and support their recovery.

DETAILED DESCRIPTION:
Cancer is a disease caused by the uncontrolled proliferation of cells in a certain part of the body and the spread of these cells. Cancer, the incidence of which is increasing, affects the patient and his family physically, psychologically, socially and spiritually, and the symptoms experienced reduce the quality of life. Breast cancer is the most common cancer in women. Tumorous tissue is removed by mastectomy, one of the breast cancer treatment methods, but individuals are exposed to physiological, psychological and social problems. It has been revealed in the literature that the education given before surgery prepares patients for surgery, reduces anxiety, accelerates the treatment process, and reduces the use of analgesia. Özberksoy et al. (2009) stated that preoperative education given to breast cancer patients reduced their postoperative pain and anxiety levels.Yutmaz (2018) stated that the video-assisted training given before mastectomy reduced pain levels on the tenth postoperative day and increased comfort. Marize et al. (2018) found that as a result of the education applied to patients who were planned for breast cancer surgery, their anxiety levels decreased and their knowledge about treatment increased. Bozdemir (2021) states that the training given to women with breast cancer after surgery is effective in preventing lymphedema and increasing the quality of life. In our study, it is aimed to examine the effect of structured education to be given to patients who are planned for mastectomy on the quality of early postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Having a mastectomy operation
* At least primary school graduate
* No psychiatric illness
* No communication problems
* Willingness to participate in the research
* Complete the data collection forms

Exclusion Criteria:

* Existence of a situation that prevents communication
* Unwillingness to participate in the research
* Incomplete answers to the questionnaire
* Individuals who are unwilling to continue the research will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
quality of recovery rate | 6 months
  The quality of recovery of patients given structured education

IPD SHARING:
Plan to Share IPD: No